CLINICAL TRIAL: NCT05984277
Title: A Phase III, Two-Arm, Parallel, Randomized, Multi-Center, Open-Label, Global Study to Determine the Efficacy of Volrustomig (MEDI5752) Plus Chemotherapy Versus Pembrolizumab Plus Chemotherapy for First-Line Treatment of Patients With Metastatic Non-Small Cell Lung Cancer (mNSCLC).
Brief Title: A Global Study of Volrustomig (MEDI5752) Plus Chemotherapy Versus Pembrolizumab Plus Chemotherapy for Participants With Metastatic Non-small Cell Lung Cancer.
Acronym: eVOLVE-Lung02
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D798AC00001; 2023-000056-38 (EudraCT Number)
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Non-small Cell Lung Cancer
Keywords: metastatic non-small cell lung cancer; non-squamous tumors; squamous tumors; PD-L1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Carboplatin; Paclitaxel; Pemetrexed

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Volrustomig plus histology-specific chemotherapy (carboplatin plus either pemetrexed or paclitaxel) via iv infusion
  Interventions: Drug: Volrustomig; Drug: Carboplatin; Drug: Paclitaxel; Drug: Pemetrexed
- Arm 2 (Active Comparator): Pembrolizumab plus histology-specific chemotherapy (carboplatin plus either pemetrexed or paclitaxel) via iv infusion
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Pemetrexed

INTERVENTIONS:
Drug: Volrustomig — Volrustomig
  Arms: Arm 1
Drug: Pembrolizumab — Pembrolizumab
  Arms: Arm 2
Drug: Carboplatin — Carboplatin
Drug: Paclitaxel — Paclitaxel
Drug: Pemetrexed — Pemetrexed

SUMMARY:
The purpose of eVOLVE-Lung02 is to test the effectiveness (efficacy) and measure the safety of volrustomig in combination with chemotherapy compared with pembrolizumab in combination with chemotherapy as 1L treatment in participants with mNSCLC in PD-L1 < 50%.

DETAILED DESCRIPTION:
Adult patients with a histologically or cytologically documented metastatic NSCLC, with tumors that lack activating EGFR, ALK, and ROS1 alterations are eligible for enrollment. Patients will be randomized in a 1:1 ratio to receive treatment with volrustomig + chemotherapy or pembrolizumab + chemotherapy. Tumor evaluation scans will be performed until disease progression as efficacy assessment. All patients will be followed for survival until the end of the study. An data monitoring committee (DMC) composed of independent experts will be convened to confirm the safety and tolerability of the proposed dose and schedule.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically documented squamous or non-squamous NSCLC.
* Stage IV NSCLC (according to Version 8 of the IASLC Staging Manual in Thoracic Oncology 2016), not amenable to curative surgery or radiation.
* Absence of sensitizing EGFR mutations and ALK and ROS1 rearrangements.
* Absence of documented tumor genomic alteration results from tests conducted as part of standard local practice in any other actionable driver oncogenes for which there are locally approved targeted first-line therapies.

Key Exclusion Criteria:

* Mixed small-cell lung cancer and NSCLC histology or sarcomatoid variant. Rare subtypes are excluded.
* Spinal cord compression.
* Symptomatic brain metastases. Brain metastases may be treated or untreated, but participants must be asymptomatic and off steroids for at least 14 days prior to start of study intervention. A minimum of 2 weeks must have elapsed between the end of brain radiotherapy and study enrollment.
* History of another primary malignancy except for:

  1. Malignancy treated with curative intent with no known active disease ≥ 2 years before the first dose of study intervention and of low potential risk for recurrence.
  2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  3. Adequately treated carcinoma in situ without evidence of disease.
* As judged by the investigator, any condition that would interfere with evaluation of the study intervention or interpretation of participant safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2028-04-24 (Estimated); Study Completion 2029-03-23 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) (using BICR assessments according to RECIST 1.1) | Up to approximately 6 years
  PFS is defined as the time from randomization until radiological progression per RECIST 1.1 as assessed by BICR, or death due to any cause (in the absence of progression), in PD-L1-negative participants.
Overall Survival (OS), in PD-L1-negative participants. | Up to approximately 6 years
  OS is defined as the time from randomization until the date of death due to any cause, in PD-L1-negative participants.

SECONDARY OUTCOMES:
PFS (using BICR assessments according to RECIST 1.1) | Up to approximately 6 years
  PFS is defined as the time from randomization until radiological progression per RECIST 1.1 as assessed by BICR, or death due to any cause (in the absence of progression). The analysis will include all randomized participants.
OS | Up to approximately 6 years
  OS is defined as the time from randomization until the date of death due to any cause. The analysis will include all randomized participants.
PFS (using Investigator assessments according to RECIST 1.1) | Up to approximately 6 years
  PFS is defined as the time from randomization until radiological progression per RECIST 1.1 as assessed by investigator, or death due to any cause (in the absence of progression).
Overall Response Rate (ORR) | Up to approximately 6 years
  ORR is defined as the proportion of participants who have a confirmed CR or confirmed PR, as determined by BICR assessments using RECIST 1.1.
Duration of Response (DoR) | Up to approximately 6 years
  DoR is defined as the time from the date of first documented response until the date of documented progression per BICR assessments using RECIST 1.1 or death due to any cause (in the absence of progression). These analyses will include participants who have a confirmed response.
PFS2 | Up to approximately 6 years
  PFS2 is defined as the time from randomization until the earliest of the progression event (following the initial investigator-assessed progression) after the start of the first subsequent therapy, or death. The date of second progression will be recorded by the investigator in the eCRF and defined according to local standard clinical practice.
Concentration of volrustomig in serum and PK parameters | Up to approximately 6 years
  To assess the PK of volrustomig
Presence of ADAs against volrustomig in serum | Up to approximately 6 years
  To investigate the immunogenicity of volrustomig.
Time-To-Deterioration (TTD) in physical functioning | Up to approximately 6 years
  To assess participant-reported physical functioning in participants treated with volrustomig plus chemotherapy and pembrolizumab plus chemotherapy.
TTD of lung cancer symptoms | Up to approximately 6 years
  To assess participant-reported pulmonary symptoms of mNSCLC in participants treated with volrustomig plus chemotherapy and pembrolizumab plus chemotherapy.

CONTACTS AND LOCATIONS:
Locations (225):
- United States (39):
  - Research Site, Prescott, Arizona
  - Research Site, Hot Springs, Arkansas
  - Research Site, Springdale, Arkansas
  - Research Site, Long Beach, California
  - Research Site, Lone Tree, Colorado
  - Research Site, Fort Myers, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Orlando, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Silver Spring, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Grand Island, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Albuquerque, New Mexico
  - Research Site, East Syracuse, New York
  - Research Site, Fresh Meadows, New York
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Horsham, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Irving, Texas
  - Research Site, Lancaster, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Tacoma, Washington
- Argentina (4):
  - Research Site, CABA
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Rosario
- Australia (5):
  - Research Site, Clayton
  - Research Site, Fitzroy
  - Research Site, Heidelberg
  - Research Site, South Brisbane
  - Research Site, Sydney
- Austria (2):
  - Research Site, Linz
  - Research Site, Wels
- Belgium (3):
  - Research Site, Aalst
  - Research Site, Antwerp
  - Research Site, Ghent
- Brazil (9):
  - Research Site, Barretos
  - Research Site, Curitiba
  - Research Site, Florianópolis
  - Research Site, Fortaleza
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Santa Cruz do Sul
  - Research Site, São Paulo
- Canada (10):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, Halifax, Nova Scotia
  - Research Site, Barrie, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Lévis, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Chicoutimi
- China (23):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Lanzhou
  - Research Site, Linhai
  - Research Site, Linyi
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shenzhen
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yangzhou
  - Research Site, Zhengzhou
- Czechia (3):
  - Research Site, Olomouc
  - Research Site, Ostrava - Vitkovice
  - Research Site, Prague
- France (15):
  - Research Site, Angers
  - Research Site, Avignon
  - Research Site, Bayonne
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Quimper
  - Research Site, Reims
  - Research Site, St-Malo
  - Research Site, Strasbourg
  - Research Site, Suresnes
  - Research Site, Toulon Naval
- Germany (17):
  - Research Site, Berlin-Zehlendorf
  - Research Site, Bonn
  - Research Site, Braunschweig
  - Research Site, Dresden
  - Research Site, Freiburg im Breisgau
  - Research Site, Gauting
  - Research Site, Georgsmarienhütte
  - Research Site, Gütersloh
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Immenhausen
  - Research Site, Koblenz
  - Research Site, Ludwigsburg
  - Research Site, Nuremberg
  - Research Site, Tübingen
  - Research Site, Velbert
- Hungary (8):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gyöngyös
  - Research Site, Gyöngyös - Mátraháza
  - Research Site, Győr
  - Research Site, Pécs
  - Research Site, Szekszárd
  - Research Site, Törökbálint
- India (7):
  - Research Site, Bengaluru
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Mysuru
  - Research Site, Nagpur
  - Research Site, Nashik
  - Research Site, Varanasi
- Italy (8):
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Ravenna
  - Research Site, Roma
- Japan (15):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Kashiwa
  - Research Site, Kawasaki-shi
  - Research Site, Kōtoku
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Sagamihara-shi
  - Research Site, Sakai
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Ube-shi
  - Research Site, Yokohama
- Netherlands (4):
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Nieuwegein
  - Research Site, Tilburg
- Poland (5):
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Przemyśl
  - Research Site, Radom
  - Research Site, Warsaw
- Slovakia (4):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Trnava
- South Africa (7):
  - Research Site, eManzimtoti
  - Research Site, George
  - Research Site, Johannesburg
  - Research Site, Pietermaritzburg
  - Research Site, Pretoria
  - Research Site, Rondebosch
  - Research Site, Soweto
- South Korea (6):
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Incheon
  - Research Site, Jinju
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (6):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Bilbao (Vizcaya)
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Palma
- Taiwan (6):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
  - Research Site, Yunlin
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Dusit
  - Research Site, Lampang
  - Research Site, Muang
  - Research Site, Songkhla
- Turkey (Türkiye) (8):
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Çankaya
  - Research Site, Diyarbakır
  - Research Site, Fatih-Istanbul
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Pamukkale
- United Kingdom (6):
  - Research Site, Birmingham
  - Research Site, Blackpool
  - Research Site, Bury St Edmunds
  - Research Site, Colchester
  - Research Site, London
  - Research Site, Truro

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. SignedData Sharing Agreement (non-negotiable contract for data accessors) must be inplace before accessing requested information. Additionally, all users will need toaccept the terms and conditions of the SAS MSE to gain access. For additionaldetails, please review the Disclosure Statements athttps://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CTIS structured data update — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D798AC00001&attachmentIdentifier=2b0100f7-99dd-4c7e-97dd-c32af12549d1&fileName=D798AC00001_CTIS_structured_data_update.pdf&versionIdentifier=